CLINICAL TRIAL: NCT05090917
Title: Development of Growth Curves in Cockayne Syndrome Type 1 and Type 2
Brief Title: Growth Curves in Cockayne Syndrome Type 1 and Type 2
Acronym: Curves-CS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7886
Record Dates: First submitted 2021-10-11; First posted 2021-10-25 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-10

CONDITIONS: Cockayne Syndrome, Type I and II
Keywords: Cockayne Syndrome; Cockayne Syndrome, Type I and II; Growth curves
MeSH Terms: conditions — Cockayne Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the natural progression of Cockayne's syndrome, affected patients also present with variable neurological and gastrointestinal damage (gastroesophageal reflux, recurrent vomiting, swallowing disorders, etc.) with varying repercussions on their growth. Acute intercurrent events such as seizures, constipation, infections can also interact with their metabolism, food intake and influence their growth. The nutritional deficit potentially involved in this growth retardation can be responsible for many manifestations such as anemia, bone fractures, fatigue, coagulation disorders responsible in total for the reduction in quality and life expectancy.

Faced with growth retardation in patients with Cockayne syndrome, medical management is difficult to establish. Is this delay part of the natural course of the pathology?

ELIGIBILITY:
Inclusion criteria:

* Minor patient
* Cockayne syndrome with molecular confirmation, treated between 01/01/1985 and 01/03/2020
* Collection of at least one growth data (height, weight, head circumference) for a given age
* Clinic compatible with type 1 or 2 Cockayne syndrome
* Holder of parental authority not opposing, after information, the reuse of their child's medical data for the purposes of this scientific research.

Exclusion criteria:

* Refusal to participate in the study.
* Lack of molecular confirmation of Cockayne syndrome
* Lack of growth data for a given age.
* Clinic not compatible with type 1 or 2 Cockayne syndrome. Exclusion of type 3 Cockayne syndromes, trichothiodystrophy and xeroderma-pigmentosum.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor patient with cockayne syndrome with molecular confirmation, treated between 01/01/1985 and 01/03/2020
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Development of growth curves in Cockayne syndrome type 1 and type 2 from existing medical data | Files analysed retrospectively from January 01, 1985 to March 01, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LAUGEL, MD, PhD, Principal Investigator — Service de Pédiatrie1 - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Pédiatrie1 - Hôpitaux Universitaires de Strasbourg, Strasbourg, France